CLINICAL TRIAL: NCT06868628
Title: A Phase 2a Study to Evaluate Microglial Activation, Safety, and Clinical Effects of Foralumab Nasal in Patients With Multiple System Atrophy (MSA)
Brief Title: A Phase 2a Study of Foralumab Nasal in Patients With Multiple System Atrophy (MSA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tiziana Life Sciences LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025P000259
Record Dates: First submitted 2025-03-06; First posted 2025-03-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Foralumab Nasal (Experimental): This study includes a 6-month observational lead-in phase followed by a 6-month open-label treatment phase with Foralumab Nasal.
  Interventions: Drug: Foralumab Nasal

INTERVENTIONS:
Drug: Foralumab Nasal — Foralumab is an anti-CD3 monoclonal antibody administered as a nasal spray. Participants will complete eight 3-week dosing cycles over the study. During each cycle, Foralumab will be administered intranasally three times per week for the first two weeks, with no administration in the third week.

SUMMARY:
A Phase 2a Study of Foralumab Nasal in Patients with Multiple System Atrophy (MSA)

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a clinical diagnosis of Clinically Established or Clinically Probable Multiple System Atrophy in accordance with 2022 MDS diagnostic criteria.
* Age 30 to 85 years, at the time of signing the informed consent.
* Stable dopaminergic treatment for at least 4 weeks before enrollment.
* Adequate hematologic parameters without ongoing transfusion support: Hemoglobin (Hb) ≥ 9 g/dL; Platelets ≥ 100 x 109 cells/L.
* Creatinine ≤ 1.5 x the upper limit of normal (ULN), or calculated creatinine clearance ≥ 60 mL/minute x 1.73 m2 per the Cockcroft-Gault formula.
* Total bilirubin ≤ 2 times the upper limit of normal (ULN) unless due to Gilbert's disease.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN.
* QT interval corrected for rate (QTcF) ≤ 470 msec for women and ≤ 450 msec for men on the ECG obtained at Screening.
* Negative urine pregnancy test within 7 days prior to the first dose of study therapy for women of child-bearing potential (WCBP), defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses any time in the preceding 24 consecutive months). Sexually active WCBP and male patients must agree to use highly effective methods to avoid pregnancy (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study and for 90 days after the completion of study treatment.
* Patients whose immunizations are fully up to date at the Screening, according to the assessment of their primary care physician and neurologist.
* Ability to provide written informed consent.

Exclusion Criteria:

* Diagnosis or suspicion of other cause for Parkinsonism or a known alternate neurologic diagnosis.
* Female patient who is pregnant, lactating, breastfeeding, or planning to become pregnant during study.
* Individuals with claustrophobia who cannot tolerate the study procedures
* Non-MRI-compatible implanted devices.
* Low-affinity binders for translocator protein (TSPO) PET ligands.
* Systemic corticosteroid treatment in the past four weeks (excluding nasal or local treatment).
* Individuals with significant cognitive impairment (i.e., MoCA score less than or equal to 20).
* Brain MRI indicative of significant abnormalities that interfere with PET-MRI co-registration (i.e., large prior hemorrhage or multiple infarcts).
* Serious cardiac condition within the last 6 months, such as uncontrolled arrhythmia, myocardial infarction, unstable angina, or heart disease defined by the New York Heart Association (NYHA) Class III or Class IV or hereditary long QT syndrome.
* Concomitant medication(s) that may cause QTc prolongation or induce Torsades de Pointes, except for antimicrobials that are used as standard of care to prevent or treat infections and other such drugs that are considered by the Investigator to be essential for patient care.
* Patients who test positive for human immunodeficiency virus (HIV), hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) or positive Epstein-Barr virus (EBV) IgM at the Screening Visit.
* Past medical history of a hematologic or solid malignancy.
* Treatment with chronic immunosuppressives such as interferon, glatiramer acetate, fingolimod, Siponimod, dimethyl fumarate, or natalizumab within the past 90 days.
* Inability to tolerate nasally administered medications.
* Nasal corticosteroids, nasal antihistamines, nasal flu dosing within the past 30 days, or anticipated need during the study.
* Chronic rhinitis, deviated septum, nasal polyps, history of sinusitis treated within the past 8 months.
* Inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, primary Sjögren's Syndrome, asthma, or type 1 diabetes.
* Neutropenia or an absolute neutrophil count of < 1,000 cells/mL or other indicators of severe immunosuppression.
* Severe lymphopenia or an absolute lymphocyte count of < 500 cells/mL
* Patients with a history of gadolinium allergy.
* A recent clinically significant active infection requiring treatment with antibiotics or other anti-infective agents within the past 15 days.
* Any other medical or surgical intervention or other condition which, in the opinion of the Principal Investigator, could compromise adherence to study requirements or confound the interpretation of study results.
* Unable or unwilling to comply with protocol requirements.
* Active COVID-19 disease.
* COVID-19 vaccine within past 10 days or any other vaccine within past 7 days (at dosing).

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from Screening to Month 6 in the total MDS-UMSARS score | From Screening to Month 6
Change in TSPO activity as measured by [F-18]PBR06 retention calculated over whole brain and within key regions of interest (ROIs) at 6 months as compared to screening | From Screening to Month 6

SECONDARY OUTCOMES:
Change from Screening to Month 6 in MDS-UMSARS Part III (motor examination) score | From Screening to Month 6
Proportion of patients with ≥30% improvement in MDS-UMSARS total score at Month 6 | From Screening to Month 6
Change from Screening to Month 6 in COMPASS-31 total score | From Screening to Month 6
Change from Screening to Month 6 in MSA-QoL summary index score | From Screening to Month 6
Percent whole brain volume change (PWBVC) between screening and 6 months | From Screening to Month 6
Percent putamen volume change (PPVC) between screening and 6 months | From Screening to Month 6
Percent cerebellar volume change (PCVC) between screening and 6 months | From Screening to Month 6
Percent pontine volume change (PPoVC) between screening and 6 months | From Screening to Month 6
Percent midbrain volume change (PMVC) between screening and 6 months | From Screening to Month 6

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wenning GK, Stankovic I, Vignatelli L, Fanciulli A, Calandra-Buonaura G, Seppi K, Palma JA, Meissner WG, Krismer F, Berg D, Cortelli P, Freeman R, Halliday G, Hoglinger G, Lang A, Ling H, Litvan I, Low P, Miki Y, Panicker J, Pellecchia MT, Quinn N, Sakakibara R, Stamelou M, Tolosa E, Tsuji S, Warner T, Poewe W, Kaufmann H. The Movement Disorder Society Criteria for the Diagnosis of Multiple System Atrophy. Mov Disord. 2022 Jun;37(6):1131-1148. doi: 10.1002/mds.29005. Epub 2022 Apr 21. PMID 35445419
- [Background] Singhal T, Cicero S, Rissanen E, Ficke J, Kukreja P, Vaquerano S, Glanz B, Dubey S, Sticka W, Seaver K, Kijewski M, Callen AM, Chu R, Carter K, Silbersweig D, Chitnis T, Bakshi R, Weiner HL. Glial Activity Load on PET Reveals Persistent "Smoldering" Inflammation in MS Despite Disease-Modifying Treatment: 18 F-PBR06 Study. Clin Nucl Med. 2024 Jun 1;49(6):491-499. doi: 10.1097/RLU.0000000000005201. Epub 2024 Apr 17. PMID 38630948
- [Background] Singhal T, O'Connor K, Dubey S, Pan H, Chu R, Hurwitz S, Cicero S, Tauhid S, Silbersweig D, Stern E, Kijewski M, DiCarli M, Weiner HL, Bakshi R. Gray matter microglial activation in relapsing vs progressive MS: A [F-18]PBR06-PET study. Neurol Neuroimmunol Neuroinflamm. 2019 Jul 1;6(5):e587. doi: 10.1212/NXI.0000000000000587. eCollection 2019 Sep. PMID 31355321
- [Background] Shahnawaz M, Mukherjee A, Pritzkow S, Mendez N, Rabadia P, Liu X, Hu B, Schmeichel A, Singer W, Wu G, Tsai AL, Shirani H, Nilsson KPR, Low PA, Soto C. Discriminating alpha-synuclein strains in Parkinson's disease and multiple system atrophy. Nature. 2020 Feb;578(7794):273-277. doi: 10.1038/s41586-020-1984-7. Epub 2020 Feb 5. PMID 32025029
- [Background] Owen DR, Yeo AJ, Gunn RN, Song K, Wadsworth G, Lewis A, Rhodes C, Pulford DJ, Bennacef I, Parker CA, StJean PL, Cardon LR, Mooser VE, Matthews PM, Rabiner EA, Rubio JP. An 18-kDa translocator protein (TSPO) polymorphism explains differences in binding affinity of the PET radioligand PBR28. J Cereb Blood Flow Metab. 2012 Jan;32(1):1-5. doi: 10.1038/jcbfm.2011.147. Epub 2011 Oct 19. PMID 22008728
- [Background] Ndayisaba A, Pitaro AT, Willett AS, Jones KA, de Gusmao CM, Olsen AL, Kim J, Rissanen E, Woods JK, Srinivasan SR, Nagy A, Nagy A, Mesidor M, Cicero S, Patel V, Oakley DH, Tuncali I, Taglieri-Noble K, Clark EC, Paulson J, Krolewski RC, Ho GP, Hung AY, Wills AM, Hayes MT, Macmore JP, Warren L, Bower PG, Langer CB, Kellerman LR, Humphreys CW, Glanz BI, Dielubanza EJ, Frosch MP, Freeman RL, Gibbons CH, Stefanova N, Chitnis T, Weiner HL, Scherzer CR, Scholz SW, Vuzman D, Cox LM, Wenning G, Schmahmann JD, Gupta AS, Novak P, Young GS, Feany MB, Singhal T, Khurana V. Clinical Trial-Ready Patient Cohorts for Multiple System Atrophy: Coupling Biospecimen and iPSC Banking to Longitudinal Deep-Phenotyping. Cerebellum. 2024 Feb;23(1):31-51. doi: 10.1007/s12311-022-01471-8. Epub 2022 Oct 3. PMID 36190676
- [Background] Moreira TG, Matos KTF, De Paula GS, Santana TMM, Da Mata RG, Pansera FC, Cortina AS, Spinola MG, Baecher-Allan CM, Keppeke GD, Jacob J, Palejwala V, Chen K, Izzy S, Healey BC, Rezende RM, Dedivitis RA, Shailubhai K, Weiner HL. Nasal Administration of Anti-CD3 Monoclonal Antibody (Foralumab) Reduces Lung Inflammation and Blood Inflammatory Biomarkers in Mild to Moderate COVID-19 Patients: A Pilot Study. Front Immunol. 2021 Aug 12;12:709861. doi: 10.3389/fimmu.2021.709861. eCollection 2021. PMID 34475873
- [Background] Meissner WG, Remy P, Giordana C, Maltete D, Derkinderen P, Houeto JL, Anheim M, Benatru I, Boraud T, Brefel-Courbon C, Carriere N, Catala H, Colin O, Corvol JC, Damier P, Dellapina E, Devos D, Drapier S, Fabbri M, Ferrier V, Foubert-Samier A, Frismand-Kryloff S, Georget A, Germain C, Grimaldi S, Hardy C, Hopes L, Krystkowiak P, Laurens B, Lefaucheur R, Mariani LL, Marques A, Marse C, Ory-Magne F, Rigalleau V, Salhi H, Saubion A, Stott SRW, Thalamas C, Thiriez C, Tir M, Wyse RK, Benard A, Rascol O; LIXIPARK Study Group. Trial of Lixisenatide in Early Parkinson's Disease. N Engl J Med. 2024 Apr 4;390(13):1176-1185. doi: 10.1056/NEJMoa2312323. PMID 38598572
- [Background] Lopes JR, Zhang X, Mayrink J, Tatematsu BK, Guo L, LeServe DS, Abou-El-Hassan H, Rong F, Dalton MJ, Oliveira MG, Lanser TB, Liu L, Butovsky O, Rezende RM, Weiner HL. Nasal administration of anti-CD3 monoclonal antibody ameliorates disease in a mouse model of Alzheimer's disease. Proc Natl Acad Sci U S A. 2023 Sep 12;120(37):e2309221120. doi: 10.1073/pnas.2309221120. Epub 2023 Sep 5. PMID 37669383
- [Background] Lavisse S, Goutal S, Wimberley C, Tonietto M, Bottlaender M, Gervais P, Kuhnast B, Peyronneau MA, Barret O, Lagarde J, Sarazin M, Hantraye P, Thiriez C, Remy P. Increased microglial activation in patients with Parkinson disease using [18F]-DPA714 TSPO PET imaging. Parkinsonism Relat Disord. 2021 Jan;82:29-36. doi: 10.1016/j.parkreldis.2020.11.011. Epub 2020 Nov 17. PMID 33242662
- [Background] Kuzkina A, Bargar C, Schmitt D, Rossle J, Wang W, Schubert AL, Tatsuoka C, Gunzler SA, Zou WQ, Volkmann J, Sommer C, Doppler K, Chen SG. Diagnostic value of skin RT-QuIC in Parkinson's disease: a two-laboratory study. NPJ Parkinsons Dis. 2021 Nov 15;7(1):99. doi: 10.1038/s41531-021-00242-2. PMID 34782640
- [Background] Jucaite A, Cselenyi Z, Kreisl WC, Rabiner EA, Varrone A, Carson RE, Rinne JO, Savage A, Schou M, Johnstrom P, Svenningsson P, Rascol O, Meissner WG, Barone P, Seppi K, Kaufmann H, Wenning GK, Poewe W, Farde L. Glia Imaging Differentiates Multiple System Atrophy from Parkinson's Disease: A Positron Emission Tomography Study with [11 C]PBR28 and Machine Learning Analysis. Mov Disord. 2022 Jan;37(1):119-129. doi: 10.1002/mds.28814. Epub 2021 Oct 5. PMID 34609758
- [Background] Ishizawa K, Komori T, Sasaki S, Arai N, Mizutani T, Hirose T. Microglial activation parallels system degeneration in multiple system atrophy. J Neuropathol Exp Neurol. 2004 Jan;63(1):43-52. doi: 10.1093/jnen/63.1.43. PMID 14748560
- [Background] Gilman S, Wenning GK, Low PA, Brooks DJ, Mathias CJ, Trojanowski JQ, Wood NW, Colosimo C, Durr A, Fowler CJ, Kaufmann H, Klockgether T, Lees A, Poewe W, Quinn N, Revesz T, Robertson D, Sandroni P, Seppi K, Vidailhet M. Second consensus statement on the diagnosis of multiple system atrophy. Neurology. 2008 Aug 26;71(9):670-6. doi: 10.1212/01.wnl.0000324625.00404.15. PMID 18725592
- [Background] Fujimura Y, Zoghbi SS, Simeon FG, Taku A, Pike VW, Innis RB, Fujita M. Quantification of translocator protein (18 kDa) in the human brain with PET and a novel radioligand, (18)F-PBR06. J Nucl Med. 2009 Jul;50(7):1047-53. doi: 10.2967/jnumed.108.060186. Epub 2009 Jun 12. PMID 19525468
- [Background] Chitnis T, Kaskow BJ, Case J, Hanus K, Li Z, Varghese JF, Healy BC, Gauthier C, Saraceno TJ, Saxena S, Lokhande H, Moreira TG, Zurawski J, Roditi RE, Bergmark RW, Giovannoni F, Torti MF, Li Z, Quintana F, Clementi WA, Shailubhai K, Weiner HL, Baecher-Allan CM. Nasal administration of anti-CD3 monoclonal antibody modulates effector CD8+ T cell function and induces a regulatory response in T cells in human subjects. Front Immunol. 2022 Nov 23;13:956907. doi: 10.3389/fimmu.2022.956907. eCollection 2022. PMID 36505477
- [Background] Chatenoud L, Bluestone JA. CD3-specific antibodies: a portal to the treatment of autoimmunity. Nat Rev Immunol. 2007 Aug;7(8):622-32. doi: 10.1038/nri2134. Epub 2007 Jul 20. PMID 17641665
- [Background] Brochard V, Combadiere B, Prigent A, Laouar Y, Perrin A, Beray-Berthat V, Bonduelle O, Alvarez-Fischer D, Callebert J, Launay JM, Duyckaerts C, Flavell RA, Hirsch EC, Hunot S. Infiltration of CD4+ lymphocytes into the brain contributes to neurodegeneration in a mouse model of Parkinson disease. J Clin Invest. 2009 Jan;119(1):182-92. doi: 10.1172/JCI36470. Epub 2008 Dec 22. PMID 19104149